CLINICAL TRIAL: NCT06300905
Title: Clinical Investigation on Oral Malodor for a New Formula of Stannous Toothpaste as Compared to Colgate Cavity Protection Toothpaste Using Organoleptic Method
Brief Title: Clinical Study on Malodor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO-2023-05-OMO-SNA-YPZ
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Oral Malodor
Keywords: Organoleptic method; oral malodor
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Brushing twice daily in the morning and evening with 2 minutes each time
  Interventions: Drug: test product; Drug: Control product
- Group II (Active Comparator): Brushing twice daily in the morning and evening with 2 minutes each time
  Interventions: Drug: test product; Drug: Control product

INTERVENTIONS:
Drug: test product — toothpaste containing 0.45% stannous fluoride
Drug: Control product — toothpaste containing 0.76% sodium monofluorophosphate

SUMMARY:
This 3-week clinical study was designed to investigate the clinical efficacy on oral malodor of a 0.454% stannous fluoride toothpaste with nitrate and pyrophosphate (referred to as SNAP) compared to Colgate Cavity Protection Toothpaste containing 0.76% sodium monofluorophosphate 12 hours post-brushing after 3 weeks of product use.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female 18 to 70 years of age
* Must be in good general health
* Must be in good oral health based on self-assessment
* Must be available during the weeks of this study for all appointment time points
* Should have a minimum of 20 natural uncrowned teeth (excluding third molars)
* Should have a baseline mean oral malodor score greater than or equal to 6.0 and less than or equal to 8.0
* Must give written informed consent
* No known history of allergy to personal care/consumer products or their ingredients

Exclusion Criteria:

* Participation in any other oral clinical studies for the duration of this study
* Full or partial (upper or lower) dentures
* Pregnant or lactating (breast feeding)
* Use of tobacco products
* History of allergy to common toothpaste ingredients
* Use of phenolic flavored products, such as mint flavored candies and chewing gum, the morning of the study and during the sampling periods
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
* Individuals who, due to medical conditions, cannot go without eating or drinking for the post use treatment evaluation time points (6 hrs. + overnight)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Organoleptic Oral Malodor Evaluations | Oral malodor evaluations at baseline & 3 weeks
  The measured levels of oral malodor will be expressed in organoleptic scales (1-9)

CONTACTS AND LOCATIONS:
Overall Officials: Deyu Hu, DDS,MS, Principal Investigator — West China Dental Institute of Chengdu
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No